CLINICAL TRIAL: NCT02652975
Title: Anticancer Treatment of Breast Cancer Related to Cardiotoxicity and Dysfunctional Endothelium
Acronym: ABCDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ABCDE_AUH
Record Dates: First submitted 2015-12-14; First posted 2016-01-12 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasms; Endothelial Dysfunction; Cardiovascular Disease; Metabolic Syndrome
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases; Metabolic Syndrome | interventions — Blood Pressure; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Category 1 (Experimental): Examination of participants prior to chemotherapy. Venous occlusion plethysmography SphygmoCor 24hour blood pressure DEXA scan Laboratory blood samples
  Interventions: Procedure: Venous occlusion plethysmography; Procedure: SphygmoCor; Procedure: 24hour blood pressure; Procedure: DEXA scan; Biological: Laboratory blood samples
- Category 2 (Experimental): Examination of participants immediately after chemotherapy. Venous occlusion plethysmography SphygmoCor 24hour blood pressure DEXA scan Laboratory blood samples
  Interventions: Procedure: Venous occlusion plethysmography; Procedure: SphygmoCor; Procedure: 24hour blood pressure; Procedure: DEXA scan; Biological: Laboratory blood samples
- Category 3 (Experimental): Examination of participants one year after chemotherapy. Venous occlusion plethysmography SphygmoCor 24hour blood pressure DEXA scan Laboratory blood samples
  Interventions: Procedure: Venous occlusion plethysmography; Procedure: SphygmoCor; Procedure: 24hour blood pressure; Procedure: DEXA scan; Biological: Laboratory blood samples

INTERVENTIONS:
Procedure: Venous occlusion plethysmography — To characterize endothelial function in vivo the effect of vasodilatating substances is measured in the forearm circuit. The substances is administered via a thin catheter placed in the Brachial artery near the elbow in local anesthesia. Once the vessels dilate, the blood flow in the forearm will increase and the flow change is a measure of the vasodilatory capacity of that substance. The change is measured with classical venous occlusion plethysmography. The method described is established at Aarhus University Hospital and has been used for several decades to illustrate the effect of vasoactive drugs on the human circulation, meaning it is a proven and well documented method.
Procedure: SphygmoCor — Applanation tonometry (pulse wave velocity and central blood pressure/arterial stiffness): The central blood pressure and the augmentation index is estimated from the shape of the radial pulse wave measured with a tonometer.
  Pulse wave velocity (PWV) is calculated from the average difference between the pulse pressure wave measured with a tonometer and the R in an ECG recorded simultaneously.
Procedure: 24hour blood pressure — 24 hour blood pressure measurement
Procedure: DEXA scan — Measurements of body composition: Total body fat and fat free mass is measured by Dual Energy X-ray Absorptiometry (DEXA).
Biological: Laboratory blood samples — Fasting blood tests are drawn from an antecubital placed catheter (albumin, ALAT/ASAT, alkaline phosphatase, bilirubin, gammaglutamyl transferase, coagulation factors, red and white blood cells, creatinin, potassium, sodium, fasting lipids, fasting glucose, hemoglobin A1C, insulin, sex hormones, von Willebrand factor, low grade inflammation markers, DNA and RNA for later analyses, including relevant coding genes).
  Further more urine samples to determine possible systemic impact of cardiovascular disease.
  We will create a biobank containing urine and blood samples from participants for future research, provided that the participant gives her permission.
  Responsibility for the biobank lies with the project responsible physician, Anders Bonde Jensen.

SUMMARY:
Several cytotoxic regimens are related to endothelial cell damage and vascular toxicity. Endothelial dysfunction is implicated in the pathogenesis of all known cardiovascular diseases (CVD) and closely related to the metabolic syndrome. Both CVD and diabetes contributes importantly to total mortality and to breast cancer (BC) specific mortality.

In the epidemiological part of the project, the investigators will determine the prevalence and incidence of cardiovascular and metabolic morbidity/mortality in early BC patients compared to the Danish background population.

In the clinical part, the investigators will study the changes of endothelial function and metabolic parameters in BC patients receiving chemotherapy.

With increasing number of BC survivors, long-term consequences of curative cancer treatment should be studied. The investigators hypothesize that cytotoxic therapy worsens metabolic parameters possibly through endothelial dysfunction. If this is true, the next step will be to evaluate how strict metabolic control will affect prognosis.

DETAILED DESCRIPTION:
1. Background

   During the past 30 years, survival of breast cancer patients has improved substantially due to earlier diagnosis, improved surgical techniques, introduction of new combination of chemotherapy, new hormonal treatment, introduction of targeted treatment, and refinement of radiation techniques. With increasing number of cancer survivors, which in part are reached by more aggressive treatment, more attention is presently being drawn to long-term consequences of curative cancer treatment.

   Comorbidity among breast cancer patients has been thoroughly studied over the past years. Previous research has however, primarily focused on prevalence of comorbidity at the time of the cancer diagnosis (manifest comorbidity) and less attention has been paid to studying latent comorbidity developing after the diagnosis, which can be a result of the treatment. Furthermore it is not known if the incidence of this later developed comorbidity is different in breast cancer patients compared to the general population. Additionally, most studies do not address specific diseases but focus on comorbidity as such. Emerging evidence, however, indicates that cardiovascular disease (CVD) (encompassing cerebrovascular disease manifested by stroke and TCI and coronary heart disease manifested by infarction, arrhythmias, heart failure and sudden death) and diabetes may play a pivotal role, because it contributes importantly both to total mortality and to breast cancer specific mortality among breast cancer survivors.

   Comorbidity at breast cancer diagnosis is an independent adverse prognostic factor. In Denmark, comorbidity was present in 26% of breast cancer patients diagnosed 2006-2008, and the presence of comorbidity increased the risk of dying from breast cancer as well as from other causes with adjusted hazard ratios for all-cause mortality of 1.45 and breast cancer-specific mortality 1.30. Most studies have, however, used a summary measure of comorbidity such as the Charlson Comorbidity Index Score, and only few studies have assessed the individual effects of specific comorbidities on the mortality among breast cancer patients. These few studies universally demonstrate that CVD and diabetes are associated with decreased overall survival. Thus, Patnaik et al showed that among breast cancer patients, women with the following comorbidities were more likely to die as a result of other causes: CVD (59.2%), COPD (52.2%), diabetes (47.8%) and previous cancer (43.8%) Fully adjusted relative hazards of the effects of comorbidities on breast cancer-specific mortality was 1.24 for CVD and 1.10 for diabetes, and among the total study population of breast cancer patients, CVD was the primary cause of death (15.9%), followed closely by breast cancer (15.1%). In a meta-analysis of studies of overall survival in breast cancer patients with preexisting diabetes, Barone et al found that preexisting diabetes was associated with an increased mortality with a hazard rate (HR) of 1.61; (95% CI, 1.46-1.78).

   Metabolic syndrome (MS) is a cluster of disorders including hypertension, type II diabetes, dyslipidemia and obesity, and certain aspects of the MS are well described in relation to breast cancer. It has been shown that obesity is associated with an increased risk of developing breast cancer among postmenopausal women, obese patients present with more advanced cancers, and women who are overweight or obese at the time of breast cancer diagnosis or gain weight after diagnosis are at increased risk of cancer recurrence and death compared with leaner women. One study have shown that the effects of adjuvant therapy is less in obese breast cancer patients. An association between diabetes and breast cancer has also been observed. Other components of the MS, including low HDL-cholesterol, high triglycerides, hypertension, and serum testosterone are, however, less well described, but may be associated with an increased breast cancer risk and a worse breast cancer prognosis. A recent study showed that patients with MS present with more aggressive tumors. In patients with metastatic disease, response to chemotherapy appears to be inferior when the patient is diagnosed with MS, as well. Emerging evidence suggest that the MS may be quite prevalent among patients with breast cancer.

   In our study the metabolic syndrome will be defined in accordance with the definition of the National Cholesterol Education Program (NCEP)/Adult Treatment Panel III (ATPIII). A diabetic FPG level is defined as FPG >7 mmol/l; impaired fasting glycemia is defined as FPG between 6.1 and 7.0 mmol/l according to World Health Organization criteria.

   Endothelial cells line the internal lumen of all the vasculature and serve as an interface between circulating blood and vascular smooth muscle cells (VSMCs). Apart from being the key participant during the process of angiogenesis, these dynamic structures can actively regulate basal vascular tone and vascular reactivity in physiological and pathological conditions. They respond to mechanical forces and neurohumoral mediators by releasing a variety of relaxing and contracting factors such as nitric oxide (NO) and prostacyclin. The balance between the vasodilatation and vasoconstriction is maintained by the endothelium, and the disruption of this balance leads to endothelial dysfunction and causes damage to the arterial wall. Endothelial cells are also responsible for the maintenance of blood fluidity and restoration of vessel wall integrity (when injured) to avoid bleeding. Endothelial cell-derived factors are also critical mediators of VSMC growth and inflammation.

   Several cytotoxic regimens have been shown to cause endothelial cell damage and vascular toxicity by various mechanisms. Thus, anthracyclines and taxanes (which forms the cornerstone of breast cancer treatment) together with cytotoxics as alkylating agents, bleomycin, vinca alkaloids and antimetabolites have been associated with endothelial cell apoptosis, oxidative stress, inflammation, coagulation disorders/thrombotic state, endothelial cell proliferation-migration, effects on VEGF, and impaired endothelial-dependent vasodilation in vitro and in vivo, although the exact mechanisms are not known. Changes in endothelial function hasten the development of micro- and macro-angiopathy and endothelial dysfunction is an important surrogate marker of atherosclerotic activity. Endothelial dysfunction has been implicated in the pathogenesis and clinical course of all known cardiovascular diseases and is associated with future risk of adverse cardiovascular events.

   Endothelial dysfunction is closely related to the MS, and a deficiency of endothelial-derived NO is believed to be the primary defect that links insulin resistance and endothelial dysfunction. It is not known whether worsening of endothelial dysfunction aggravates elements of the MS.
2. Objective

The aim of this research program is to study the changes of endothelial function and metabolic parameters in patients receiving chemotherapy for early stage breast cancer, and to compare these parameters with healthy age matched controls.

Our theory is that cytotoxic therapy can induce endothelial cell damage and vascular toxicity causing endothelial dysfunction. The investigators believe that endothelial dysfunction is a mediator in the MS and predisposes to later cardiovascular disease, thus rendering patients receiving cytotoxic therapy at risk of these conditions.

The investigators hypothesize that:

1. Cytotoxic therapy induces endothelial dysfunction in predisposed early breast cancer patients.
2. Metabolic syndrome may be aggravated by cytotoxic therapy, possibly through worsening of endothelial dysfunction.
3. Treatment of early breast cancer (chemotherapy, antihormonal therapy and/or trastuzumab) aggravates preexisting CVD and/or metabolic disease and may induce the metabolic syndrome.

3) Methods

The study is a clinical case-control study with the inclusion of 90 patients divided into 3 groups as stated below. 30 healthy women with the same age will participate as controls (group 4).

Group 1: Newly diagnosed patients with early breast cancer. Investigated immediately prior to start of adjuvant therapy.

Group 2: Early breast cancer patients, who have received standard treatment. Investigated immediately after completion of adjuvant chemotherapy.

Group 3: Early breast cancer patients, who have received standard treatment. Investigated 1 year after completed chemotherapy.

Group 4: Healthy, age-matched controls. Controls will be recruited from an internet resource (www.forsoegsperson.dk):

The test program will consist of the following investigations:

1. To characterize endothelial function in vivo the effect of vasodilatating substances is measured in the forearm circuit. The substances is administered via a thin catheter placed in the Brachial artery near the elbow in local anesthesia. Once the vessels dilate, the blood flow in the forearm will increase and the flow change is a measure of the vasodilatory capacity of that substance. The change is measured with classical venous occlusion plethysmography. The method described is established at Aarhus University Hospital and has been used for several decades to illustrate the effect of vasoactive drugs on the human circulation, meaning it is a proven and well documented method.
2. Applanation tonometry (pulse wave velocity and central blood pressure/arterial stiffness): The central blood pressure and the augmentation index is estimated from the shape of the radial pulse wave measured with a tonometer.

   Pulse wave velocity (PWV) is calculated from the average difference between the pulse pressure wave measured with a tonometer and the R in an ECG recorded simultaneously.
3. Medical history: A full medical history including use of medication is obtained from every subject. Age, smoking status and concurrent medication. For patients tumor characteristics and anticancer treatment will also be described.
4. Clinical examination: A regular objective examination is performed including weight, height (BMI) and measurements of hip and waist circumference.
5. Measurements of body composition: Total body fat and fat free mass is measured by Dual Energy X-ray Absorptiometry (DEXA).
6. Electrocardiography: A conventional 12 lead surface electrocardiogram is recorded.
7. 24 hour blood pressure measurement
8. Laboratory tests: Fasting blood tests are drawn from an antecubital placed catheter (albumin, ALAT/ASAT, alkaline phosphatase, bilirubin, gammaglutamyl transferase, coagulation factors, red and white blood cells, creatinin, potassium, sodium, fasting lipids, fasting glucose, hemoglobin A1C, insulin, sex hormones, von Willebrand factor, low grade inflammation markers, DNA and RNA for later analyses, including relevant coding genes).

   Further more urine samples to determine possible systemic impact of cardiovascular disease.

   The investigators will create a biobank containing urine and blood samples from participants for future research, provided that the participant gives her permission.

   Responsibility for the biobank lies with the project responsible physician, Anders Bonde Jensen.
9. To characterize the overall risk of cardiovascular death within 10 years, the investigators will use a well- established and validated method called SCORE using age, gender, smoking status, systolic blood pressure and plasma cholesterol for risk stratification.
10. Every premenopausal woman will be asked about the possibility of her being pregnant. In case of doubt the investigators will do a pregnancy test (urine hcg)

ELIGIBILITY:
Inclusion Criteria:

* women referred to receive adjuvant chemotherapy for primary operable non-metastatic breast cancer

Exclusion Criteria:

* former og actual use of cytostatics
* pregnancy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial dysfunction evaluated using plethysmography. | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
Changes in aortic pressure evaluated using applanation tonometry (SphygmoCor) | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
Changes in blood pressure evaluated by 24 hour blood pressure measurements. | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
Changes in metabolic measurements using the blood samples listed in descriptive field. | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
  P-Kolesterol, P-Kolesterol HDL, P-Kolesterol LDL, P-Triglyceride, P-Glukose, P-Progesteron, P-Testosteron, P-Von Willebrand-faktor, P-Natrium, P-Kalium, P-Kreatinin and P-Østradiol.
Changes in body composition using DEXA scans | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
Changes in risk of cardiovascular death within 10 years using the SCORE-system. | Measured before start of chemotherapy (week 0), immediately after ended chemotherapy (week 18) and one year after ended chemotherapy (week 70).
  The SCORE-system is a well- established and validated method using age, gender, smoking status, systolic blood pressure and plasma cholesterol for risk stratification.

CONTACTS AND LOCATIONS:
Overall Officials: Anders B. Jensen, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fredslund SO, Gravholt CH, Laursen BE, Jensen AB. Key metabolic parameters change significantly in early breast cancer survivors: an explorative PILOT study. J Transl Med. 2019 Apr 1;17(1):105. doi: 10.1186/s12967-019-1850-2. PMID 30935397